CLINICAL TRIAL: NCT05730855
Title: Diagnostic Accuracy of lncRNA DQ786243 and miRNA146a in Saliva of Oral Potentially Malignant Lesions
Status: Completed | Type: Observational
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Salsabeel, Lecturer, Fayoum University
Other Study IDs: 1152014
Record Dates: First submitted 2023-02-07; First posted 2023-02-16 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Potentially Malignant Lesions; Oral Lichen Planus; Leukoplakia, Oral
Keywords: lncRNA DQ786243; saliva; oral potentially malignant lesions; miRNA146a
MeSH Terms: conditions — Lichen Planus, Oral; Leukoplakia, Oral

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Oral Lichen Planus
  Interventions: Diagnostic Test: Real-time Polymerase Chain Reaction technique
- Leukoplakia
  Interventions: Diagnostic Test: Real-time Polymerase Chain Reaction technique
- Healthy control
  Interventions: Diagnostic Test: Real-time Polymerase Chain Reaction technique

INTERVENTIONS:
Diagnostic Test: Real-time Polymerase Chain Reaction technique — Real-time Polymerase Chain Reaction technique

SUMMARY:
The aim of this study is to evaluate salivary expression of lncRNA DQ786243 as a potential marker for diagnosis of oral potentially malignant lesions compared to normal controls and its effect on salivary expression of miRNA146a.

ELIGIBILITY:
Inclusion Criteria:

* participants will be divided into 3 groups:

Group I: patients suffering from oral lichen planus Group II: patients suffering from leukoplakia Group III: healthy subjects who are systemically free, non-smokers, and not suffering from any oral mucosal lesions.

Exclusion Criteria:

* Subjects taking any drugs inducing any changes that could affect the salivary flow.
* Pregnant females.
* Subjects have any allergies, infectious diseases or active dental abscesses during one month before saliva sampling.
* Patients receiving any drugs related to the oral lesions in the past 6 month prior to sample collection.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Egyptian Population
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2022-12-24 (Actual); Study Completion 2023-01-23 (Actual)

PRIMARY OUTCOMES:
salivary expression of lncDQ786243 in OLP, Leukoplakia, control | 2 months

SECONDARY OUTCOMES:
salivary expression of miRNA146a in OLP, Leukoplakia, control | 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Fayoum University, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP